CLINICAL TRIAL: NCT03301558
Title: The Effect of Sodium Bicarbonate (Nephrotrans®) on Calcification Propensity of Serum in Kidney Transplant Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study not started due to organizational reasons
Sponsor: Prim. Priv. Doz. Dr. Daniel Cejka (Other)
Collaborators: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Sponsor-Investigator, Prim. Priv. Doz. Dr. Daniel Cejka, Head of Nephrology, Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KTR-Bic-T50
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to either receive low-dose (1500 mg/d) sodium bicarbonate followed by high-dose (3000mg/d) sodium bicarbonate (sequence A-B) or to receive high-dose sodium bicarbonate followed by low-dose sodium bicarbonate (sequence B-A) with washout-phases in between.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose sodium bicarbonate (Active Comparator): Low dose 1500 mg sodium bicarbonate (Nephrotrans®) per day (500mg tablets 3x/day) for 14 ± 3 days. The patients will be advised to take one capsule with breakfast, one with lunch and one with dinner (schedule 1-1-1).
  Interventions: Drug: Low dose sodium bicarbonate
- High Dose sodium bicarbonate (Active Comparator): High dose 3000 mg of sodium bicarbonate (Nephrotrans®) per day (500mg tablets 3x/day) for 14 ± 3 days. The patients will be advised to take two capsules with breakfast, two with lunch and two with dinner (schedule 2-2-2).
  Interventions: Drug: High dose sodium bicarbonate

INTERVENTIONS:
Drug: Low dose sodium bicarbonate — 1500 mg sodium bicarbonate
  Other Names: Nephrotrans
  Arms: Low dose sodium bicarbonate
Drug: High dose sodium bicarbonate — 3000 mg sodium bicarbonate
  Other Names: Nephrotrans
  Arms: High Dose sodium bicarbonate

SUMMARY:
This is a single-center, prospective, open-label, randomized, cross-over study.

DETAILED DESCRIPTION:
The primary hypothesis (H1) is that the T50 value will change between wash-out and high-dose (3000mg/d) sodium bicarbonate (Nephrotrans®) substitution.

The 0-hypothesis (H0) is that substitution of 3000 mg/d sodium bicarbonate (Nephrotrans®) has no effect on T50-values as compared to wash-out-phase.

Patients will be randomized in a 1:1 ratio to either receive low-dose (1500 mg/d) sodium bicarbonate followed by high-dose (3000mg/d) sodium bicarbonate (sequence A-B) or to receive high-dose sodium bicarbonate followed by low-dose sodium bicarbonate (sequence B-A) with washout-phases in between.

Patients will be randomized in a 1:1 ratio to either receive low-dose (1500 mg/d) sodium bicarbonate followed by high-dose (3000mg/d) sodium bicarbonate (sequence A-B) or to receive high-dose sodium bicarbonate followed by low-dose sodium bicarbonate (sequence B-A) with washout-phases in between. The study will start with an initial run-in wash-out phase, where all sodium bicarbonate or other alkalizing treatment taken by the patient as standard of care will be discontinued. Consequently, there will be a sodium bicarbonate treatment (high dose/low dose) phase, followed by a wash-out phase, followed by another sodium bicarbonate treatment (high dose/low dose) phase, followed by a final wash-out phase. Each study phase, including wash-out phases as well as low-dose and high-dose treatment phases will be 14 ±3 days of duration. Patients will be followed up to 12weeks after randomization until the last study visit of the final wash-out phase.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Prevalent (≥ 6 months after kidney transplantation) kidney transplant recipients
* eGFR (CKD-EPI formula) between 10 and 50 ml/min/1.73 m²
* Patient has provided informed consent prior to initiation of any study related procedure

Exclusion Criteria:

* Allergy to sodium bicarbonate or any component of Nephrotrans®, namely soy or peanuts (reported cross-reactivity to peanuts has been reported in patients with soy-allergy).
* Unstable clinical condition (e.g. uncontrolled heart failure, clinical uremia, uncontrolled hypertension, impending initiation of dialysis treatment…) as judged by the recruiting physician
* Pregnant and nursing (lactating) women
* Unwillingness to discontinue current medication with sodium bicarbonate
* Unwillingness to discontinue antacids containing aluminum, calcium carbonate, magnesium, lactate, citrate, bicarbonate or mixtures thereof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Propensity of serum for calcification | 12 weeks
  The primary outcome is change in the mean T50 values between different study phases (treatment vs. control).

SECONDARY OUTCOMES:
Serum bicarbonate levels | 12 weeks
  The secondary outcome is change of serum bicarbonate levels between different study phases.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cejka, MD, Principal Investigator — Head of Nephrology
Locations (1):
- Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No